CLINICAL TRIAL: NCT07279792
Title: Implications of Post-Operative Irrigation Fluid's Osmolarity on the Recurrence of Non-Muscle Invasive Bladder Cancer Following Transurethral Resection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS 685/2024
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-09

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer; Nonmuscle Invasive Bladder Cancer; Irrigation; Hypertonic Saline; Normal Saline; Distilled Water
MeSH Terms: conditions — Neoplasms | interventions — Saline Solution; Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous Bladder Irrigation with distilled water (Active Comparator)
  Interventions: Drug: Continuous Bladder Irrigation with distilled water
- Continuous Bladder Irrigation with normal saline (Active Comparator)
  Interventions: Drug: Continuous Bladder Irrigation with normal saline
- Continuous Bladder Irrigation with hypertonic saline (Active Comparator)
  Interventions: Drug: Continuous Bladder Irrigation with hypertonic saline

INTERVENTIONS:
Drug: Continuous Bladder Irrigation with distilled water — Continuous Bladder Irrigation with distilled water post non muscle invasive bladder cancer urethral resection by endoscopy
  Arms: Continuous Bladder Irrigation with distilled water
Drug: Continuous Bladder Irrigation with normal saline — Continuous Bladder Irrigation with normal saline post non muscle invasive bladder cancer urethral resection by endoscopy
  Arms: Continuous Bladder Irrigation with normal saline
Drug: Continuous Bladder Irrigation with hypertonic saline — Continuous Bladder Irrigation with hypertonic saline post non muscle invasive bladder cancer urethral resection by endoscopy
  Arms: Continuous Bladder Irrigation with hypertonic saline

SUMMARY:
This randomized controlled trial will evaluate the efficacy of three bladder irrigation solutions - distilled water (DW), normal saline (NS), and hypertonic saline (HS) - as continuous bladder irrigation (CBI) following transurethral resection of non-muscle invasive bladder cancer (NMIBC). Short term (6 months) recurrence and progression free survival are mainly evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients of non-muscle invasive urinary bladder urothelial carcinoma amenable for complete resection

Exclusion Criteria:

* Patients with post-operative complications that need prolonged irrigation.
* Patient who underwent incomplete resection during TURBT.
* When large bladder perforation was suspected during TURBT.
* Patients with chronic kidney disease.
* Muscle invasive disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Risk of Recurrence | 6 months
Risk of progression of bladder cancer | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes